CLINICAL TRIAL: NCT00819507
Title: Effects of a Novel Formulation of Fluocinonide 0.1% Cream on Skin Barrier Function in Atopic Dermatitis
Brief Title: VANOS Cream and Skin Barrier Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Principal Investigator, Eric Simpson, Professor, Dermatology, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4590
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Atopic Dermatitis
Keywords: Skin barrier; Atopic Dermatitis; Corticosteroid; Effects on skin severity and barrier function
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Fluocinonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vanos Cream (Experimental): glucocorticoid cream
  Interventions: Drug: Fluocinonide

INTERVENTIONS:
Drug: Fluocinonide — Fluocinonide 0.1% cream topical daily for two weeks

SUMMARY:
The purpose of this study is to determine the effect of short-term therapy using "VANOS Cream," a super-potent topical steroid cream on skin barrier function in patients with atopic dermatitis. This cream is already approved for this indication, but the investigators will further examine its effects on the skin barrier. This cream is a novel formulation of fluocinonide designed to enhance compliance with a cream base, but have the skin barrier repair properties of an ointment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD according to Hanifin-Rajka criteria (see Appendix B)
* Age 12 years or older
* Must have an Investigator's Global Assessment (IGA) Score of Moderate, Severe, or Very Severe (See Appendix C)
* Must have failed to achieve adequate disease despite adequate topical or systemic therapy
* Must be a candidate, according to the principal investigator and standard of care, for a super-potent topical steroid course. Subjects that are candidates for super-potent topical steroids are defined as subjects whose disease is not adequately controlled with medium-potency topical steroids or systemic therapy, including phototherapy.

Exclusion Criteria:

* Active skin infection
* Hypersensitivity to any ingredients in Vanos cream
* Previous use of super-potent topical steroids within 2 weeks of starting study (Class I steroid).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University Department of Dermatology, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vanos Cream
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vanos Cream
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 39 [17 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, Non-Hispanic | 19
  African-American | 2
  Asian | 2
  Hispanic | 1
  Mixed race | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Eczema Severity and Area Index
Description: The eczema area and severity index (EAS I) is a validated composite score measuring physical signs of atopic dermatitis. The scale ranges from 0-72. The components measuring severity are four signs/symptoms of atopic dermatitis: erythema, population, excoriation and lichenification on a scale of 0-3 for each body of the four body regions (head/neck, trunk, arms, legs). The component measuring area is a body surface area measurement of each region. The area and severity of each body region is weighted based on size of region which are added together for the complete score. The score for each patient's with scores between 0 and 7 are considered mild ,between 7 and 21 are considered moderate, and greater than 21 are considered severe. In this study the change in EASI score between baseline and end of study (baseline EASI subtracted from end of study EASI) was calculated as a final outcome data point.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Vanos Cream
Number analyzed (Participants) | 25
units | 6.01 (7.9)
Statistical Analysis 1: Comparison: Vanos Cream; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 6.01

2. Secondary Outcome: Change in Transepidermal Water Loss
Description: A measure of water flux out the skin using a small non-invasive probe. Values can range between 0-no water loss and over 100-severe water loss. This measure indicates the degree of skin barrier permeability with lower values indicating lower permeability (improved skin barrier function).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: G/m^2/hr
Arm/Group | Vanos Cream
Number analyzed (Participants) | 25
G/m^2/hr | 14.35 (16)
Statistical Analysis 1: Comparison: Vanos Cream; Test type: Superiority; p < 0.01, t-test, 2 sided; Median Difference (Final Values) = 14.35

ADVERSE EVENTS:
Arm/Group | Vanos Cream
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vanos Cream (N=25)
burning (Skin and subcutaneous tissue disorders) | 1 (1) — burning for 2 days, rated as mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No